CLINICAL TRIAL: NCT03418922
Title: A Phase 1b Trial of Lenvatinib Plus Nivolumab in Subjects With Hepatocellular Carcinoma
Brief Title: A Study of Lenvatinib Plus Nivolumab in Participants With Hepatocellular Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: E7080-J081-117
Record Dates: First submitted 2018-01-26; First posted 2018-02-01 (Actual); Results first posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2022-05

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib; Nivolumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 1: Lenvatinib Plus Nivolumab (Experimental): Participants will receive specified doses of lenvatinib (oral) and nivolumab (intravenous) on specified days.
  Interventions: Drug: Lenvatinib; Drug: Nivolumab
- Part 2: Lenvatinib Plus Nivolumab (Experimental): If tolerable in Part 1, participants will receive specified doses of lenvatinib and nivolumab on specified days until criteria for discontinuation are met.
  Interventions: Drug: Lenvatinib; Drug: Nivolumab

INTERVENTIONS:
Drug: Lenvatinib — Specified doses will be administered orally on specified days.
Drug: Nivolumab — Specified doses will be administered intravenously on specified days.

SUMMARY:
The primary objective of this study is to evaluate the tolerability and safety of a combination of lenvatinib plus nivolumab in participants with hepatocellular carcinoma (HCC).

ELIGIBILITY:
Inclusion Criteria:

* Participants must have confirmed diagnosis of hepatocellular carcinoma (HCC) with any of the following criteria:

  * Histologically or cytologically confirmed diagnosis of HCC, excluding fibrolamellar, sarcomatoid or mixed cholangio-HCC tumors
  * Clinically confirmed diagnosis of HCC according to American Association for the Study of Liver Diseases criteria, including cirrhosis of any etiology and/or chronic hepatitis B or C infection
* Part 1: HCC for which no other appropriate therapy is available; Part 2: No prior systemic therapy for advanced/unresectable HCC
* Participants categorized to stage B (not applicable for transarterial chemoembolization), or stage C based on Barcelona Clinic Liver Cancer staging system
* Child-Pugh score A
* Participants must have an Eastern Cooperative Oncology Group Performance Status of 0 to 1
* Age greater than or equal to (>=) 20 years at the time of informed consent

Exclusion Criteria:

* Active co-infection with hepatitis B and hepatitis C
* Participants with any active, known, or suspected autoimmune disease
* Participants being treated with drugs that strongly inhibit or induce CYP3A4 and that may be possibly used during this study
* Females who are breastfeeding or pregnant

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-01-16 (Actual); Primary Completion 2022-12-28 (Actual); Study Completion 2022-12-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- Japan (6):
  - Eisai Trial Site 1, Kashiwa, Chiba
  - Eisai Trial Site 6, Iizuka, Fukuoka
  - Eisai Trial Site 3, Kawasaki, Kanagawa
  - Eisai Trial Site 4, Sayama, Osaka
  - Eisai Trial Site 2, Chuo-ku, Tokyo
  - Eisai Trial Site 5, Chiba

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in two parts (Part 1 and Part 2) between 16 January 2018 and 28 December 2022 at 1 site for Part 1 and 6 sites for Part 2 in Japan.
Pre-assignment Details: A total of 30 participants were enrolled and received treatment. Of these, 6 participants were enrolled in Part 1 and 24 were enrolled in the Part 2.
Groups:
- Part 1: Lenvatinib 12 mg or 8 mg + Nivolumab 240 mg: In Part 1, Participants received lenvatinib 12 mg or 8 mg capsules, orally, once daily, in combination with nivolumab 240 mg, infusion, intravenously, Q2W on Days 1 and 15 of each 28 days cycle. Participants with body weight greater than or equal to (>=) 60 kg received lenvatinib 12 mg and participants with body weight less than (<) 60 kg, received lenvatinib 8 mg.
- Part 2: Lenvatinib 12 mg or 8 mg + Nivolumab 240 mg: In Part 2, participants received lenvatinib 12 mg or 8 mg capsules, orally, once daily, in combination with nivolumab 240 mg, infusion, intravenously, Q2W on Days 1 and 15 of each 28 days Cycle. Participants with body weight >=60 kg received lenvatinib 12 mg, participants with body weight <60 kg, received lenvatinib 8 mg.
Period: Overall Study
Arm/Group | Part 1: Lenvatinib 12 mg or 8 mg + Nivolumab 240 mg | Part 2: Lenvatinib 12 mg or 8 mg + Nivolumab 240 mg
Started | 6 | 24
Completed | 4 | 18
Not Completed | 2 | 6
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Adverse Event | 2 | 2
Not completed — Death | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received at least 1 dose of lenvatinib or nivolumab.
Groups:
- Part 1: Lenvatinib 12 mg or 8 mg + Nivolumab 240 mg: In Part 1, Participants received lenvatinib 12 mg or 8 mg capsules, orally, once daily, in combination with nivolumab 240 mg, infusion, intravenously, Q2W on Days 1 and 15 of each 28 days cycle. Participants with body weight >=60 kg received lenvatinib 12 mg and participants with body weight less than <60 kg, received lenvatinib 8 mg.
- Total: Total of all reporting groups
Arm/Group | Part 1: Lenvatinib 12 mg or 8 mg + Nivolumab 240 mg | Part 2: Lenvatinib 12 mg or 8 mg + Nivolumab 240 mg | Total
Number analyzed (Participants) | 6 | 24 | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.5 (1.87) | 67.1 (10.74) | 68.4 (9.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 6
  Male | 5 | 19 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 6 | 23 | 29
  Chinese | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Dose-Limiting Toxicities (DLTs)
Description: DLT was graded according to Common Terminology Criteria for Adverse Events version 4.03 (CTCAE v4.03). DLT was defined as any of the following hematological or non-hematological toxicities considered to be at least possibly related to lenvatinib and/or nivolumab occurring during Cycle 1: 1) Febrile neutropenia or Grade 4 neutropenia for >7 days; 2) Grade 4 thrombocytopenia and Grade 3 thrombocytopenia with bleeding; 3) Grade 4 anemia; 4) Clinical deterioration manifested by drug-related hepatic decompensation; 5) >=Grade 3 non-hematological laboratory abnormalities with clinical symptoms that persisted; 6) Other Grade 3 toxicity lasting >3 days or Grade 4 non-hematological toxicity of any duration; 7) Grade 2 uveitis, eye pain, or blurred vision that did not respond to topical therapy; 8) Failure to administer 8 or more dose of the planned administration number of study drug in Cycle 1 as a result of treatment-related toxicity.
Time Frame: Cycle 1 (Cycle length = 28 days)
Population: The DLT analysis set included all participants who had completed Cycle 1 without major protocol deviation with at least 75 percent (%) of study drug compliance and at least 2 doses of nivolumab and were assessed for DLT, and participants who had experienced DLT during Cycle 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Lenvatinib 12 mg or 8 mg + Nivolumab 240 mg
Number analyzed (Participants) | 6
Participants | 0

2. Primary Outcome: Part 1 and Part 2: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: A TEAE was defined as an adverse event (AE) that emerged during treatment and until the 30 days after the last dose or until the participants initiated new anticancer therapy, whichever was earlier, was absent at pretreatment (Baseline) or reemerged during treatment, was present at pretreatment (Baseline) but stopped before treatment, or worsened in severity during treatment relative to the pretreatment state, when the AE was continuous. An SAE was any untoward medical occurrence that at any dose: resulted in death, was life-threatening (that is, participant was at immediate risk of death from AE as it occurred; this did not include an event that, had it occurred in a more severe form or was allowed to continue, might have caused death), required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect (in the child of a participant who was exposed to the study drug).
Time Frame: From the first dose of study drug until 30 days after the last dose (up to 53 months)
Population: Safety analysis set included all participants who received at least 1 dose of lenvatinib or nivolumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Lenvatinib 12 mg or 8 mg + Nivolumab 240 mg | Part 2: Lenvatinib 12 mg or 8 mg + Nivolumab 240 mg
Number analyzed (Participants) | 6 | 24
Participants
  TEAEs | 6 | 24
  SAEs | 3 | 12

3. Primary Outcome: Mean Change From Baseline in Vital Sign: Weight
Description: Mean change from baseline in weight were evaluated.
Time Frame: Baseline, up to Month 53
Population: Safety analysis set included all participants who received at least 1 dose of lenvatinib or nivolumab. Here, "Overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: kilogram
Arm/Group | Part 1: Lenvatinib 12 mg or 8 mg + Nivolumab 240 mg | Part 2: Lenvatinib 12 mg or 8 mg + Nivolumab 240 mg
Number analyzed (Participants) | 6 | 23
kilogram | 2.82 (3.931) | -3.10 (4.953)

4. Primary Outcome: Mean Change From Baseline in Vital Sign: Body Mass Index
Description: Mean change from baseline in body mass index were evaluated.
Time Frame: Baseline, up to Month 53
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: kilogram per square meter
Arm/Group | Part 1: Lenvatinib 12 mg or 8 mg + Nivolumab 240 mg | Part 2: Lenvatinib 12 mg or 8 mg + Nivolumab 240 mg
Number analyzed (Participants) | 6 | 23
kilogram per square meter | 1.10 (1.434) | -1.12 (1.811)

5. Primary Outcome: Mean Change From Baseline in Vital Sign: SpO2 (Oxygen Saturation)
Description: Mean change from baseline in SpO2 were evaluated.
Time Frame: Baseline, up to Month 53
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of blood oxygen saturation
Arm/Group | Part 1: Lenvatinib 12 mg or 8 mg + Nivolumab 240 mg | Part 2: Lenvatinib 12 mg or 8 mg + Nivolumab 240 mg
Number analyzed (Participants) | 6 | 23
percentage of blood oxygen saturation | 0.2 (0.75) | -0.6 (1.41)

6. Primary Outcome: Number of Participants With Treatment-Emergent Markedly Abnormal Laboratory Values (TEMAVs)
Description: Treatment-emergent markedly abnormal laboratory value was defined as a postbaseline laboratory value with grade 3 or higher, and with a grade increase from baseline, (that is [i.e.] increasing grade 0 to 3 or higher, grade 1 to 3 or higher, grade 2 to 3 or higher, grade 3 to 4 or 5, grade 4 to 5). Test abnormalities were graded by Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 as Grade 1 =mild; Grade 2 =moderate; Grade 3/Grade 4 =severe/life-threatening, Grade 5 =death.
Time Frame: From the first dose of study drug until 30 days after the last dose (up to 53 months)
Population: Safety analysis set included all participants who received at least 1 dose of lenvatinib or nivolumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Lenvatinib 12 mg or 8 mg + Nivolumab 240 mg | Part 2: Lenvatinib 12 mg or 8 mg + Nivolumab 240 mg
Number analyzed (Participants) | 6 | 24
Participants
  Hemoglobin: Markedly Abnormal Low | 0 | 2
  Hemoglobin: Markedly Abnormal High | 0 | 0
  Platelets: Markedly Abnormal Low | 2 | 1
  Leukocytes: Markedly Abnormal Low | 0 | 0
  Leukocytes: Markedly Abnormal High | 0 | 0
  Lymphocytes: Markedly Abnormal Low | 2 | 4
  Lymphocytes: Markedly Abnormal High | 0 | 0
  Neutrophils: Markedly Abnormal Low | 0 | 3
  Prothrombin international normalized ratio: Markedly Abnormal High | 0 | 0
  Alkaline phosphatase: Markedly Abnormal High | 0 | 1
  Aspartate aminotransferase: Markedly Abnormal High | 0 | 6
  Alanine aminotransferase: Markedly Abnormal High | 1 | 1
  Gamma-glutamyl transferase: Markedly Abnormal High | 1 | 6
  Bilirubin: Markedly Abnormal High | 0 | 3
  Creatinine: Markedly Abnormal High | 1 | 0
  Glucose: Markedly Abnormal Low | 0 | 0
  Glucose: Markedly Abnormal High | 0 | 4
  Albumin: Markedly Abnormal Low | 1 | 2
  Cholesterol: Markedly Abnormal High | 0 | 0
  Triglycerides: Markedly Abnormal High | 0 | 1
  Phosphate: Markedly Abnormal Low | 0 | 3
  Sodium: Markedly Abnormal Low | 0 | 3
  Sodium: Markedly Abnormal High | 0 | 0
  Potassium: Markedly Abnormal Low | 0 | 3
  Potassium: Markedly Abnormal High | 0 | 0
  Calcium corrected: Markedly Abnormal Low | 0 | 0
  Calcium corrected: Markedly Abnormal High | 0 | 0
  Magnesium: Markedly Abnormal Low | 0 | 1
  Magnesium: Markedly Abnormal High | 0 | 0
  Amylase: Markedly Abnormal High | 1 | 1
  Lipase: Markedly Abnormal High | 3 | 5

7. Primary Outcome: Number of Participants With Highest Post-Baseline Values for Eastern Cooperative Oncology Group Performance Status (ECOG-PS) Scale
Description: Performance status assessments were based on 5-grade ECOG scale (from 0 to 4), where 0=fully active, able to carry on all pre-disease performance without restriction; 1=restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature (e.g., light house work, office work); 2=ambulatory and capable of all self-care but unable to carry out any work activities, up and about more than 50% of waking hours; 3=capable of only limited self-care, confined to bed or chair more than 50% of waking hours; 4=completely disabled, cannot carry on any self-care, totally confined to bed or chair; 5=dead.
Time Frame: Baseline, up to Month 53
Population: Safety analysis set included all participants who received at least 1 dose of lenvatinib or nivolumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Lenvatinib 12 mg or 8 mg + Nivolumab 240 mg | Part 2: Lenvatinib 12 mg or 8 mg + Nivolumab 240 mg
Number analyzed (Participants) | 6 | 24
Participants
  Grade 0 | 0 | 15
  Grade 1 | 5 | 6
  Grade 2 | 0 | 1
  Grade 3 | 1 | 2
  Grade 4 | 0 | 0

8. Primary Outcome: Change From Baseline in Left Ventricular Ejection Fraction (LVEF)
Description: Change from baseline in left ventricular ejection fraction (LVEF) were evaluated by multigated acquisition scan (MUGA) or echocardiogram.
Time Frame: Baseline, up to Month 53
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: %LVEF
Arm/Group | Part 1: Lenvatinib 12 mg or 8 mg + Nivolumab 240 mg | Part 2: Lenvatinib 12 mg or 8 mg + Nivolumab 240 mg
Number analyzed (Participants) | 5 | 19
%LVEF | 0.0 (2.00) | 0.4 (4.65)

9. Secondary Outcome: Part 1 and Part 2: Objective Response Rate (ORR) Based on Modified Response Evaluation Criteria in Solid Tumors (mRECIST) Assessed by Investigator Review
Description: ORR was defined as the percentage of participants who had best overall response (BOR) of complete response (CR) or partial response (PR) based on mRECIST assessed by investigator review. CR defined as disappearance of all target lesions and non-target lesions (a short diameter is less than 10 millimeters [mm] if it exists in a lymph node). PR defined as at least 30% decrease in the sum of diameter of all target lesions without unequivocal progression of all non-target lesions, as compared with Baseline.
Time Frame: From the first dose of study drug to the first date of documentation of PD or death, whichever occurred first (up to 52 months)
Population: Efficacy analysis set included all participants who received at least 1 dose of lenvatinib and nivolumab.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: Lenvatinib 12 mg or 8 mg + Nivolumab 240 mg | Part 2: Lenvatinib 12 mg or 8 mg + Nivolumab 240 mg
Number analyzed (Participants) | 6 | 24
percentage of participants | 66.7 [22.3 to 95.7] | 79.2 [57.8 to 92.9]

10. Secondary Outcome: Part 1, Cmax: Maximum Observed Plasma Concentration for Lenvatinib
Description: Cmax was defined as the maximum plasma concentration for lenvatinib. Cmax was derived by non-compartmental analysis using lenvatinib plasma concentrations.
Time Frame: Cycle 1 Day 1: 0-24 hours post-dose (Cycle length=28 days)
Population: Pharmacokinetic (PK) analysis set included all participants who had received at least 1 dose of lenvatinib and nivolumab, and had evaluable concentration data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- Lenvatinib 8 mg + Nivolumab 240 mg: Participants with body weight <60 kg received lenvatinib 8 mg capsules, orally, once daily, in combination with nivolumab 240 mg, infusion, intravenously, Q2W on Days 1 and 15 of each 28 days cycle.
- Lenvatinib 12 mg + Nivolumab 240 mg: Participants with body weight >=60 kg received lenvatinib 12 mg capsules, orally, once daily, in combination with nivolumab 240 mg, infusion, intravenously, Q2W on Days 1 and 15 of each 28 days cycle.
Arm/Group | Lenvatinib 8 mg + Nivolumab 240 mg | Lenvatinib 12 mg + Nivolumab 240 mg
Number analyzed (Participants) | 2 | 4
nanogram per milliliter (ng/mL) | 93.3 (16.8) | 122 (46.3)

11. Secondary Outcome: Part 1, Tmax: Time to Reach the Cmax for Lenvatinib
Description: Tmax was defined as the time to reach maximum observed plasma concentration (Cmax) for lenvatinib. Tmax was derived by non-compartmental analysis using lenvatinib plasma concentrations.
Time Frame: Cycle 1 Day 1: 0-24 hours post-dose (Cycle length=28 days)
Population: PK analysis set included all participants who had received at least 1 dose of lenvatinib and nivolumab and had evaluable concentration data.
Measure: Median (Full Range); unit: hours
Arm/Group | Lenvatinib 8 mg + Nivolumab 240 mg | Lenvatinib 12 mg + Nivolumab 240 mg
Number analyzed (Participants) | 2 | 4
hours | 1.45 [0.87 to 2.02] | 3.97 [1.80 to 7.52]

12. Secondary Outcome: Part 1, AUC(0-t): Area Under the Plasma Concentration-time Curve From Zero Time to the Last Measurable Point for Lenvatinib
Description: AUC(0-t) was defined as the area under the plasma concentration-time curve from 0 time to last measurable point for lenvatinib. AUC(0-t) was derived by non-compartmental analysis using lenvatinib plasma concentrations.
Time Frame: Cycle 1 Day 1 and Day 15: 0-24 hours post-dose (Cycle length=28 days)
Population: PK analysis set included all participants who had received at least 1 dose of lenvatinib and nivolumab and had evaluable concentration data. Here, "number analyzed" signifies participants who were evaluable for specified timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | Lenvatinib 8 mg + Nivolumab 240 mg | Lenvatinib 12 mg + Nivolumab 240 mg
Number analyzed (Participants) | 2 | 4
nanogram*hour per milliliter (ng*h/mL)
  Cycle 1 Day 1 | 882 (0.0801) | 1380 (36.0)
  Cycle 1 Day 15: number analyzed (Participants) | 2 | 3
  Cycle 1 Day 15 | 1410 (16.7) | 1920 (17.2)

13. Secondary Outcome: Part 1, AUC(0-Inf): Area Under the Plasma Concentration-time Curve From Zero to Infinity for Lenvatinib
Description: AUC(0-Inf) was defined as the area under the plasma concentration-time curve from 0 to infinity for lenvatinib. AUC(0-Inf) was derived by non-compartmental analysis using lenvatinib plasma concentrations.
Time Frame: Cycle 1 Day 1: 0-24 hours post-dose (Cycle length=28 days)
Population: PK analysis set included all participants who had received at least 1 dose of lenvatinib and nivolumab and had evaluable concentration data. Here, "Overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Lenvatinib 8 mg + Nivolumab 240 mg | Lenvatinib 12 mg + Nivolumab 240 mg
Number analyzed (Participants) | 2 | 1
ng*h/mL | 987 (6.10) | 1630 (NA) — Geometric Coefficient of Variation could not be calculated for a single participant.

14. Secondary Outcome: Part 1, t1/2: Terminal Elimination Phase Half-Life for Lenvatinib
Description: t1/2 was defined as the terminal elimination phase half-life for lenvatinib. t1/2 was derived by non-compartmental analysis using lenvatinib plasma concentrations.
Time Frame: Cycle 1 Day 1: 0-24 hours post-dose (Cycle length=28 days)
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Lenvatinib 8 mg + Nivolumab 240 mg | Lenvatinib 12 mg + Nivolumab 240 mg
Number analyzed (Participants) | 2 | 1
hours | 6.77 (27.1) | 8.95 (NA) — Geometric Coefficient of Variation could not be calculated for a single participant.

15. Secondary Outcome: Part 1, CL/F: Apparent Total Clearance for Lenvatinib
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. CL/F was calculated as (Dose/AUC(0-inf))/F. Where AUC(0-inf) is the area under the plasma concentration-time curve from zero to infinity and F is the bioavailability of the drug.
Time Frame: Cycle 1 Day 1: 0-24 hours post-dose (Cycle length=28 days)
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour (L/h)
Arm/Group | Lenvatinib 8 mg + Nivolumab 240 mg | Lenvatinib 12 mg + Nivolumab 240 mg
Number analyzed (Participants) | 2 | 1
liter per hour (L/h) | 8.09 (6.30) | 7.37 (NA) — Geometric Coefficient of Variation could not be calculated for a single participant.

16. Secondary Outcome: Part 1, Vz/F: Apparent Terminal Volume of Distribution for Lenvatinib
Description: Volume of distribution was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Vz/F was calculated as (CL/F)/Lambda Z. Where, CL/F is the apparent total clearance and lambda Z is the apparent terminal elimination rate constant.
Time Frame: Cycle 1 Day 1: 0-24 hours post-dose (Cycle length=28 days)
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter
Arm/Group | Lenvatinib 8 mg + Nivolumab 240 mg | Lenvatinib 12 mg + Nivolumab 240 mg
Number analyzed (Participants) | 2 | 1
liter | 79.0 (20.4) | 95.1 (NA) — Geometric Coefficient of Variation could not be calculated for a single participant.

17. Secondary Outcome: Part 1, Css,Max: Maximum Observed Plasma Concentration at Steady State for Lenvatinib
Description: Css,max was defined as the maximum plasma concentration at steady state for lenvatinib. Css,max was derived by non-compartmental analysis using lenvatinib plasma concentrations.
Time Frame: Cycle 1 Day 15: 0-24 hours post-dose (Cycle length=28 days)
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Lenvatinib 8 mg + Nivolumab 240 mg | Lenvatinib 12 mg + Nivolumab 240 mg
Number analyzed (Participants) | 2 | 3
ng/mL | 139 (29.5) | 164 (9.93)

18. Secondary Outcome: Part 1, Css,Min: Minimum Observed Plasma Concentration at Steady State for Lenvatinib
Description: Css,min is the minimum plasma concentration at steady state for lenvatinib. Css,min was derived by non-compartmental analysis using lenvatinib plasma concentrations.
Time Frame: Cycle 1 Day 15: 0-24 hours post-dose (Cycle length=28 days)
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Lenvatinib 8 mg + Nivolumab 240 mg | Lenvatinib 12 mg + Nivolumab 240 mg
Number analyzed (Participants) | 2 | 3
ng/mL | 13.5 (15.8) | 28.2 (48.7)

19. Secondary Outcome: Part 1, Tss,Max: Time to Maximum Observed Concentration at Steady State For Lenvatinib
Description: Tss,Max was defined as the time to reach maximum observed plasma concentration of lenvatinib at steady state. Tss,Max was derived by non-compartmental analysis using lenvatinib plasma concentrations.
Time Frame: Cycle 1 Day 15: 0-24 hours post-dose (Cycle length=28 days)
Population: as for outcome 13
Measure: Median (Full Range); unit: hours
Arm/Group | Lenvatinib 8 mg + Nivolumab 240 mg | Lenvatinib 12 mg + Nivolumab 240 mg
Number analyzed (Participants) | 2 | 3
hours | 3.94 [3.85 to 4.02] | 3.93 [3.92 to 7.98]

20. Secondary Outcome: Part 1, Rac (Cmax): Accumulation Ratio of Cmax for Lenvatinib
Description: Rac(Cmax) was calculated as Css,max at Cycle 1 Day 15/Cmax at Cycle 1 Day 1.
Time Frame: Cycle 1 Day 1 and Day 15: 0-24 hours post-dose (Cycle length=28 days)
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Lenvatinib 8 mg + Nivolumab 240 mg | Lenvatinib 12 mg + Nivolumab 240 mg
Number analyzed (Participants) | 2 | 3
ratio | 1.48 (12.4) | 1.28 (62.4)

21. Secondary Outcome: Part 1, Rac (AUC0-t): Accumulation Ratio of AUC(0-t) for Lenvatinib
Description: Rac(AUC) was calculated as AUC(0-t) at Cycle 1 Day 15/AUC(0-t) at Cycle 1 Day 1.
Time Frame: Cycle 1 Day 1 and Day 15: 0-24 hours post-dose (Cycle length=28 days)
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Groups:
- Lenvatinib 12 mg + Nivolumab 240 mgEdit: Participants with body weight >=60 kg received lenvatinib 12 mg capsules, orally, once daily, in combination with nivolumab 240 mg, infusion, intravenously, Q2W on Days 1 and 15 of each 28 days cycle.
Arm/Group | Lenvatinib 8 mg + Nivolumab 240 mg | Lenvatinib 12 mg + Nivolumab 240 mgEdit
Number analyzed (Participants) | 2 | 3
ratio | 1.59 (17.0) | 1.38 (47.1)

22. Secondary Outcome: Part 1, MRT: Mean Residence Time for Lenvatinib
Description: MRT was derived by non-compartmental analysis using lenvatinib plasma concentrations.
Time Frame: Cycle 1 Day 1: 0-24 hours post-dose (Cycle length=28 days)
Population: as for outcome 13
Measure: Median (Full Range); unit: hours
Arm/Group | Lenvatinib 8 mg + Nivolumab 240 mg | Lenvatinib 12 mg + Nivolumab 240 mg
Number analyzed (Participants) | 2 | 1
hours | 10.9 [9.35 to 12.4] | 13.7 [13.7 to 13.7]

ADVERSE EVENTS:
Time Frame: From the first dose of study drug until 30 days after the last dose (up to 53 months)
Description: The safety analysis set included all participants who had received at least 1 dose of study drug.
Arm/Group | Part 1: Lenvatinib 12 mg or 8 mg + Nivolumab 240 mg | Part 2: Lenvatinib 12 mg or 8 mg + Nivolumab 240 mg
All-Cause Mortality (participants affected / at risk) | 1/6 | 18/24
Serious Adverse Events (participants affected / at risk) | 3/6 | 12/24
Other Adverse Events (participants affected / at risk) | 6/6 | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Lenvatinib 12 mg or 8 mg + Nivolumab 240 mg (N=6) | Part 2: Lenvatinib 12 mg or 8 mg + Nivolumab 240 mg (N=24)
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Adrenocorticotropic hormone deficiency (Endocrine disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Oedema (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
C-reactive protein increased (Investigations) | 0 | 1
Hyperammonaemia (Metabolism and nutrition disorders) | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 0 | 2
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Aortic dissection (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Lenvatinib 12 mg or 8 mg + Nivolumab 240 mg (N=6) | Part 2: Lenvatinib 12 mg or 8 mg + Nivolumab 240 mg (N=24)
Anaemia (Blood and lymphatic system disorders) | 0 | 3
Eosinophilia (Blood and lymphatic system disorders) | 0 | 3
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 3 | 7
Hyperthyroidism (Endocrine disorders) | 2 | 1
Adrenocorticotropic hormone deficiency (Endocrine disorders) | 0 | 2
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Dry eye (Eye disorders) | 0 | 1
Periorbital inflammation (Eye disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 15
Stomatitis (Gastrointestinal disorders) | 2 | 8
Constipation (Gastrointestinal disorders) | 2 | 6
Nausea (Gastrointestinal disorders) | 4 | 4
Abdominal pain (Gastrointestinal disorders) | 0 | 6
Abdominal pain upper (Gastrointestinal disorders) | 0 | 4
Vomiting (Gastrointestinal disorders) | 2 | 2
Abdominal discomfort (Gastrointestinal disorders) | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 2
Periodontal disease (Gastrointestinal disorders) | 0 | 2
Anal erosion (Gastrointestinal disorders) | 0 | 1
Angular cheilitis (Gastrointestinal disorders) | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 1
Gingival pain (Gastrointestinal disorders) | 0 | 1
Glossitis (Gastrointestinal disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0
Varices oesophageal (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 5 | 4
Malaise (General disorders) | 0 | 9
Pyrexia (General disorders) | 1 | 5
Oedema peripheral (General disorders) | 1 | 4
Oedema due to hepatic disease (General disorders) | 0 | 1
Thirst (General disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 2
Cholestasis (Hepatobiliary disorders) | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1
Contrast media allergy (Immune system disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 6
Gingivitis (Infections and infestations) | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Bronchitis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Laryngitis (Infections and infestations) | 0 | 1
Liver abscess (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Scratch (Injury, poisoning and procedural complications) | 0 | 2
Face injury (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0
Weight decreased (Investigations) | 0 | 8
Aspartate aminotransferase increased (Investigations) | 1 | 4
Lipase increased (Investigations) | 2 | 2
Alanine aminotransferase increased (Investigations) | 1 | 2
Blood thyroid stimulating hormone increased (Investigations) | 0 | 3
Gamma-glutamyltransferase increased (Investigations) | 1 | 2
Ammonia increased (Investigations) | 0 | 2
Haemoglobin decreased (Investigations) | 0 | 2
Lymphocyte count decreased (Investigations) | 1 | 1
Platelet count decreased (Investigations) | 2 | 0
Amylase increased (Investigations) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1
Blood urea increased (Investigations) | 1 | 0
C-reactive protein increased (Investigations) | 0 | 1
Urinary occult blood positive (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 4 | 11
Hyperammonaemia (Metabolism and nutrition disorders) | 1 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Headache (Nervous system disorders) | 1 | 4
Dysgeusia (Nervous system disorders) | 1 | 1
Hepatic encephalopathy (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1
Taste disorder (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 0 | 1
Vagus nerve disorder (Nervous system disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 5
Proteinuria (Renal and urinary disorders) | 3 | 11
Dysuria (Renal and urinary disorders) | 0 | 1
Menstruation irregular (Reproductive system and breast disorders) | 0 | 1
Scrotal oedema (Reproductive system and breast disorders) | 1 | 0
Scrotum erosion (Reproductive system and breast disorders) | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 7
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 | 16
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 6
Rash (Skin and subcutaneous tissue disorders) | 0 | 5
Erythema (Skin and subcutaneous tissue disorders) | 1 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Lichen planus (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-02-05): https://cdn.clinicaltrials.gov/large-docs/22/NCT03418922/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-21): https://cdn.clinicaltrials.gov/large-docs/22/NCT03418922/SAP_001.pdf